CLINICAL TRIAL: NCT02099981
Title: Restoration of Retinal Vascular Responses in Type 1 Diabetic Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: Protocol 22503
Record Dates: First submitted 2014-03-26; First posted 2014-03-31 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Diabetic Retinopathy
Keywords: Diabetes; Diabetic; Retinopathy; Ophthalmology; Eye; Eyes
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Retinal Diseases | interventions — pimagedine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Experimental): Control subjects will receive AG.
  Interventions: Drug: Aminoguanidine
- Type 1 diabetes (Experimental): Type 1 diabetic subjects will receive AG.
  Interventions: Drug: Aminoguanidine

INTERVENTIONS:
Drug: Aminoguanidine
  Other Names: AG

SUMMARY:
Diabetic retinopathy is the leading cause of blindness in the developed world. The causes of the disease are poorly understood. One of the earliest changes that occur in the retinas of diabetic patients, well before overt retinopathy is observed, is a reduction in light-evoked increases in blood flow in retinal vessels. The loss of this vascular response may lead to retinal hypoxia and it has been suggested that hypoxia could be a principal cause of diabetic retinopathy.

The long-term goals of this project are to determine whether decreased blood flow in diabetic patients and the resulting retinal hypoxia contributes to the development of diabetic retinopathy and whether restoration of normal blood flow in diabetic patients slows or prevents the development of retinopathy.

DETAILED DESCRIPTION:
The immediate goal of the proposed project is to determine whether administration of aminoguanidine (AG) restores light--evoked vasodilations in the retinas of patients without advanced retinopathy. We will also determine whether AG improves contrast sensitivity in diabetic patients. The proposed experiments are as a first step in developing new therapies to prevent diabetic retinopathy.

Study participants will be asked to come to the University of Minnesota on three (3) occasions (the visits will last for up to 2, 5 and 3 hours respectively).

Visit 1. During the screening visit (first and shortest visit), consent will be obtained and baseline labs collected (Hemoglobin A1c and Creatinine). Demographic information (date of birth, gender, race), subjects characteristics (weight, height, blood pressure and pulse) and relevant medical history will be recorded.

Visit 2. Vessel dilation testing: Control and diabetic subjects will present to the Ophthalmology Research Unit at the University of Minnesota. Prior to the imaging examination, each subject will receive dilating eye drops (1% Tropicamide) to prevent accommodation of the pupil and brief eye exam will be performed. Measurement of resting vessel diameter and light--evoked vessel dilation will be made using the Imedos Systems "Dynamic Vessel Analyzer". Subjects will be instructed to look at a fixation spot and a 350 s sequence of fundus images will be acquired during baseline and stimulation period. After completion of the initial vasodilation measurements, both control and diabetic subjects will be given 150 mg AG orally and measurement of resting vessel diameter and light--evoked vasodilation will be repeated 90 minutes later.

Visit 3. Contrast sensitivity testing: Contrast sensitivity will be assessed in un-dilated control and diabetic subjects. Contrast sensitivity will be determined both before and after AG administration using a CSV-100 test chart (VectorVision) and will be measured at 3, 6, 12, and 18 cycles per degree.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes between 18 and 65 years of age
* Diabetes duration between 5 to 20 years.
* Normal report or minor findings on a dilated eye exam
* Healthy subjects on no medications

Exclusion Criteria:

Current diagnosis or history of:

* hypertension
* dyslipidemia
* epilepsy
* glaucoma or other ocular disease
* renal insufficiency/failure (creatinine >1.5 mg/dL)
* pregnancy or breastfeeding.
* smoker

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The vascular response to flicker | 90 minutes
  The vascular response will be defined as the ratio of the maximal vessel diameter observed during the stimulation period, compared to the mean diameter during the control period

SECONDARY OUTCOMES:
Contrast sensitivity | 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Seaquist, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center Fairview, Minneapolis, Minnesota, United States